CLINICAL TRIAL: NCT03262116
Title: Individualizing Automated Closed Loop Glucose Control Through Pharmacokinetic Profiling in an Insulin-Only Bionic Pancreas
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Devices are not available
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boston University (Other)
Responsible Party: Principal Investigator, Steven J. Russell, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2017P001778
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Results first posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: bionic pancreas; insulin; continuous glucose monitor; type 1 diabetes; insulin pharmacokinetics
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Insulin Lispro; Insulin; Insulin Aspart

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be blinded to the type of insulin used in the iLet bionic pancreas each arm of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Bionic Pancreas - Humalog (Experimental): Subjects will participate in one week of wearing the insulin only bionic pancreas using humalog as the rapid acting insulin.
  Interventions: Drug: Humalog; Device: Bionic Pancreas
- Bionic Pancreas - Novolog (Experimental): Subjects will participate in one week of wearing the insulin only bionic pancreas using novolog as the rapid acting insulin.
  Interventions: Drug: Novolog; Device: Bionic Pancreas
- Bionic Pancreas - BC222 insulin lispro (Experimental): Subjects will participate in one week of wearing the insulin only bionic pancreas using BC222 insulin lispro as the rapid acting insulin.
  Interventions: Drug: BC222 insulin lispro; Device: Bionic Pancreas

INTERVENTIONS:
Drug: Humalog — Subjects will participate in one week of wearing the insulin only bionic pancreas using humalog as the rapid acting insulin.
  Other Names: insulin
  Arms: Bionic Pancreas - Humalog
Drug: Novolog — Subjects will participate in one week of wearing the insulin only bionic pancreas using novolog as the rapid acting insulin.
  Other Names: insulin
  Arms: Bionic Pancreas - Novolog
Drug: BC222 insulin lispro — Subjects will participate in one week of wearing the insulin only bionic pancreas using BC222 insulin lispro as the rapid acting insulin.
  Other Names: insulin
  Arms: Bionic Pancreas - BC222 insulin lispro
Device: Bionic Pancreas — The insulin-only bionic pancreas will be used in all three arms of the study

SUMMARY:
Subjects will participate in three weeks of the bionic pancreas in the insulin-only configuration. Each week, subjects will use a different rapid acting insulin analog -- Humalog, Novolog, or BC222 insulin lispro -- in a randomized cross-over order.

DETAILED DESCRIPTION:
The investigators hypothesize that differences in the PK characteristics of insulin analogs will lead to differences in glycemic outcomes when delivered by the insulin-only configuration of the bionic pancreas. Specifically, the investigators predict that insulin analogs that have faster absorption (numerically lower Tmax and/or T½max) and insulin analogs that have faster clearance (numerically lower terminal half-life) will result in lower mean glucose and/or a lower percentage of time in the hypoglycemic range.

Up to 30 subjects will participate in three 7-day study arms using insulin lispro, insulin aspart, and BC222 lispro in the bionic pancreas in random order. The co-primary outcomes will be mean CGMG and fraction of time spent with CGMG <54 mg/dl with comparisons made between arms for individual participants. Secondary analyses will include time in glycemic ranges (<50, <60, <70, 70-120, 70-180, >180, >250 mg/dl), coefficient of variation, mean postprandial excursion (difference in CGMG from the time of meal announcement to the peak CGMG in the first 4 hours after the meal announcement) for both mixed meal challenges, number of symptomatic hypoglycemic events, grams of carbohydrate consumed to treat hypoglycemia, and TDD of insulin, between arms for individual subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and have had clinical type 1 diabetes for at least one year
* Diabetes managed using an insulin pump for ≥ 6 months
* Have used a CGM for at least one cumulative month over the last 12 months
* Prescription medication regimen stable for > 1 month (except for medications that will not affect the safety of the study and are not expected to affect any outcome of the study, in the judgment of the principal investigator)
* Willing to remain within a 250 mile radius of MGH. No air travel will be allowed, and subjects will still be expected to follow the visit schedule as described.
* Willing to wear one Dexcom CGM sensor, and one leur-lock compatible infusion set that must be replaced every other day
* Have a mobile phone they will have access to at all times during the study for making contact with study staff

Exclusion Criteria:

* Unable to provide informed consent (e.g. impaired cognition or judgment)
* Unable to safely comply with study procedures and reporting requirements (e.g. impairment of vision or dexterity that prevents safe operation of the bionic pancreas, impaired memory, unable to speak and read English)
* Current participation in another diabetes-related clinical trial that, in the judgment of the principal investigator, will compromise the results of this study or the safety of the subject
* Pregnancy (positive urine HCG), breast feeding, plan to become pregnant in the immediate future, or sexually active without use of contraception Subjects must use acceptable contraception for the two weeks prior to the study, throughout the study and for the two weeks following the study.

Acceptable contraception methods include: Oral contraceptive pill (OCP), Intrauterine Device (IUD, hormonal or copper), Male condoms, Female condoms, Diaphragm or cervical cap with spermicide, Contraceptive patch (such as OrthoEvra), Contraceptive implant (such as Implanon, Nexplanon), Vaginal ring (such as NuvaRing), Progestin shot (such as Depo-Provera), Male partner with a vasectomy proven to be effective by semen analysis

* Current alcohol abuse (intake averaging > 3 drinks daily in last 30 days) or other substance abuse (use within the last 6 months of controlled substances other than marijuana without a prescription)
* Unwilling or unable or to avoid use of drugs that may dull the sensorium, reduce sensitivity to symptoms of hypoglycemia, or hinder decision making during the period of participation in the study (use of beta blockers will be allowed as long as the dose is stable and the subject does not meet the criteria for hypoglycemia unawareness while taking that stable dose, but use of benzodiazepines or narcotics or other central nervous system depressants, even if by prescription, may be excluded according to the judgment of the principal investigator)
* Renal failure requiring dialysis
* Estimated Glomerular filtration rate <15 mL/min/1.732
* Personal history of cystic fibrosis, severe pancreatitis, pancreatic tumor, pancreatectomy or any other pancreatic disease leading to diabetes mellitus.
* Any known history of coronary artery disease including, but not limited to, history of myocardial infarction, stress test showing ischemia, history of angina, or history of intervention such as coronary artery bypass grafting, percutaneous coronary intervention, or enzymatic lysis of a presumed coronary occlusion)
* Abnormal EKG consistent with coronary artery disease or increased risk of malignant arrhythmia including, but not limited to, evidence of active ischemia, prior myocardial infarction, proximal LAD critical stenosis (Wellen's sign), prolonged QT interval (> 440 ms). Non-specific ST segment and T wave changes are not grounds for exclusion in the absence of symptoms or history of heart disease. A reassuring evaluation by a cardiologist after an abnormal EKG finding may allow participation.
* Congestive heart failure (established history of CHF, lower extremity edema, paroxysmal nocturnal dyspnea, or orthopnea)
* History of TIA or stroke15. Recent history of diabetic ketoacidosis (DKA) or severe hypoglycemia in the last 6 months. Severe hypoglycemia is defined as an event that required assistance of another person due to altered consciousness, and required another person to actively administer carbohydrate, glucagon, or other resuscitative actions. This means that the participant was impaired cognitively to the point that he/she was unable to treat himself/herself, was unable to verbalize his/ her needs, was incoherent, disoriented, and/or combative, or experienced seizure or coma.
* History of more than 1 episode of DKA requiring hospitalization in the last 2 years
* History of more than 1 episode of severe hypoglycemia in the last year.
* Untreated or inadequately treated mental illness (indicators would include symptoms such as psychosis, hallucinations, mania, and any psychiatric hospitalization in the last year), or treatment with anti-psychotic medications that are known to affect glucose regulation.
* Electrically powered implants (e.g. cochlear implants, neurostimulators) that might be susceptible to RF interference
* Unable to completely avoid acetaminophen for duration of study
* Established history of allergy or severe reaction to adhesive or tape that must be used in the study
* History of eating disorder within the last 2 years, such as anorexia, bulimia, or diabulemia or omission of insulin to manipulate weight
* History of intentional, inappropriate administration of insulin leading to severe hypoglycemia requiring treatment
* Use of oral (e.g. thiazolidinediones, biguanides, sulfonylureas, glitinides, DPP-4 inhibitors, SGLT-2 inhibitors) or non-insulin injectable (GLP-1 agonists, amylin) anti-diabetic medications
* Any diagnosed allergy to insulin lispro or insulin aspart
* Lives in or frequents areas with poor Verizon wireless network coverage (which would prevent study staff from contacting subjects)
* Any factors that, in the opinion of the principal investigator would interfere with the safe completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Russell, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 20 subjects signed the consent form and screened into the study. 2 subjects were found to be ineligible after they were enrolled. 13 pariticpants were randomized. The numbers listed here, and throughout the record only represent unique participants. Dyads, including designated contacts, are not used. No relevant data was collected from designated contacts.
Groups:
- Insulin-only Bionic Pancreas With BC222 Lispro, Then Insulin Lispro, Then Insulin Aspart; Insulin-only Bionic Pancreas With BC222 Lispro, Then Insulin Aspart, Then Insulin Lispro; Insulin-only Bionic Pancreas With Insulin Lispro, Then BC222 Lispro, Then Insulin Aspart; Insulin-only Bionic Pancreas With Insulin Lispro, Then Insulin Aspart, Then BC222 Lispro; Insulin-only Bionic Pancreas With Insulin Aspart, Then BC222 Lispro, Then Insulin Lispro; Insulin-only Bionic Pancreas With Insulin Aspart, Then Insulin Lispro, Then BC222 Lispro: Participants were randomized to complete three weeks using the insulin-only bionic pancreas. Participants would complete 7 days of each intervention in random order, including 7 days using the bionic pancreas with insulin lispro, 7 days with the bionic pancreas using insulin aspart and 7 days with the bionic pancreas using BC222 lispro. It was planned that all participants would complete all three interventions.
  The numbers listed in the participant flow, and throughout the record only represent unique participants. Dyads, including designated contacts, are not used. No data was collected from designated contacts taht is relevant to this protocol.
  The study had be terminated before all participants could complete all interventions. All available data are reported here.
Period: Overall Study
Arm/Group | Insulin-only Bionic Pancreas With BC222 Lispro, Then Insulin Lispro, Then Insulin Aspart | Insulin-only Bionic Pancreas With BC222 Lispro, Then Insulin Aspart, Then Insulin Lispro | Insulin-only Bionic Pancreas With Insulin Lispro, Then BC222 Lispro, Then Insulin Aspart | Insulin-only Bionic Pancreas With Insulin Lispro, Then Insulin Aspart, Then BC222 Lispro | Insulin-only Bionic Pancreas With Insulin Aspart, Then BC222 Lispro, Then Insulin Lispro | Insulin-only Bionic Pancreas With Insulin Aspart, Then Insulin Lispro, Then BC222 Lispro
Started | 2 | 3 | 2 | 2 | 2 | 2
Completed | 2 | 1 | 1 | 1 | 1 | 0
Not Completed | 0 | 2 | 1 | 1 | 1 | 2
Not completed — Physician Decision | 0 | 2 | 1 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: 20 participants consented to participate. 13 participants were randomized to complete three weeks using the insulin-only bionic pancreas. Only 6 completed all three arms.
  The numbers listed in the participant flow, and throughout the record only represent unique participants. Dyads, including designated contacts, are not used. No data was collected from designated contacts that is relevant to this protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin-only Bionic Pancreas With BC222 Lispro, Then Insulin Lispro, Then Insulin Aspart | Insulin-only Bionic Pancreas With BC222 Lispro, Then Insulin Aspart, Then Insulin Lispro | Insulin-only Bionic Pancreas With Insulin Lispro, Then BC222 Lispro, Then Insulin Aspart | Insulin-only Bionic Pancreas With Insulin Lispro, Then Insulin Aspart, Then BC222 Lispro | Insulin-only Bionic Pancreas With Insulin Aspart, Then BC222 Lispro, Then Insulin Lispro | Insulin-only Bionic Pancreas With Insulin Aspart, Then Insulin Lispro, Then BC222 Lispro | Total
Number analyzed (Participants) | 2 | 3 | 2 | 2 | 2 | 2 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.0 (14.1) | 40.7 (17.6) | 70.5 (14.8) | 33.0 (9.9) | 47.0 (14.1) | 50.0 (15.6) | 47.8 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 2 | 1 | 1 | 7
  Male | 2 | 1 | 1 | 0 | 1 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 2 | 3 | 2 | 2 | 1 | 2 | 12
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 2 | 2 | 2 | 2 | 13
Hemoglobin A1c [Mean (Standard Deviation); unit: percent of glycated hemoglobin] | 6.7 (0.8) | 6.9 (0.9) | 6.9 (0.2) | 6.2 (0.5) | 7.2 (0.8) | 6.4 (0.5) | 6.7 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Average Continuous Glucose Monitor (CGM) Glucose
Description: The average glucose achieved by the bionic pancreas as measured by the continuous glucose monitor during each arm
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Insulin-only Bionic Pancreas With BC222 Lispro; Insulin-only Bionic Pancreas With Insulin Lispro; Insulin-only Bionic Pancreas With Insulin Aspart: Participants were randomized to complete three weeks using the insulin-only bionic pancreas. Participants would complete 7 days of each intervention in random order, including 7 days using the bionic pancreas with insulin lispro, 7 days with the bionic pancreas using insulin aspart and 7 days with the bionic pancreas using BC222 lispro. It was planned that all participants would complete all three interventions.
  The numbers listed in the participant flow, and throughout the record only represent unique participants. Dyads, including designated contacts, are not used. No data was collected from designated contacts taht is relevant to this protocol.
  The study had be terminated before all participants could complete all interventions. All available data are reported here.
Arm/Group | Insulin-only Bionic Pancreas With BC222 Lispro | Insulin-only Bionic Pancreas With Insulin Lispro | Insulin-only Bionic Pancreas With Insulin Aspart
Number analyzed (Participants) | 8 | 8 | 8
mg/dl | 157.0 (9.2) | 151.4 (13.1) | 151.2 (13.8)

2. Primary Outcome: Percentage of Time Spent With CGM Glucose < 54 mg/dl
Description: The amount of time the subject spent in the hypoglycemic range < 54 mg/dl as measured by the continuous glucose monitor during each arm
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: percentage of CGM glucose values
Arm/Group | Insulin-only Bionic Pancreas With BC222 Lispro | Insulin-only Bionic Pancreas With Insulin Lispro | Insulin-only Bionic Pancreas With Insulin Aspart
Number analyzed (Participants) | 8 | 8 | 8
percentage of CGM glucose values | 0.30 (0.53) | 0.55 (0.26) | 1.01 (0.70)

3. Secondary Outcome: Percentage of Time Spent Within Each of the Following Ranges:
Description: The amount of time subject's spent in each of the listed glucose ranges as measured by the continuous glucose monitor during each bionic pancreas arm
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: percentage of CGM glucose values
Arm/Group | Insulin-only Bionic Pancreas With BC222 Lispro | Insulin-only Bionic Pancreas With Insulin Lispro | Insulin-only Bionic Pancreas With Insulin Aspart
Number analyzed (Participants) | 8 | 8 | 8
percentage of CGM glucose values
  % time CGM glcuose < 50 mg/dl | 0.20 (0.42) | 0.24 (0.21) | 0.63 (0.50)
  % time CGM glcuose < 60 mg/dl | 0.80 (0.88) | 1.31 (0.55) | 1.85 (1.05)
  % time CGM glcuose < 70 mg/dl | 2.65 (1.71) | 3.59 (1.71) | 4.31 (1.66)
  % time CGM glcuose 70-120 mg/dl | 27.49 (5.04) | 27.20 (5.53) | 30.44 (5.57)
  % time CGM glcuose 70-180 mg/dl | 67.77 (8.57) | 72.16 (10.34) | 70.06 (10.25)
  % time CGM glcuose >180 mg/dl | 29.58 (7.79) | 24.26 (9.29) | 25.63 (9.02)
  % time CGM glcuose > 250 mg/dl | 7.67 (3.55) | 5.21 (5.24) | 7.11 (6.41)

4. Secondary Outcome: Within Day Coefficient of Variation
Description: A measure of dispersion of glucose values around the mean
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: percentage of CGM glucose values
Arm/Group | Insulin-only Bionic Pancreas With BC222 Lispro | Insulin-only Bionic Pancreas With Insulin Lispro | Insulin-only Bionic Pancreas With Insulin Aspart
Number analyzed (Participants) | 8 | 8 | 8
percentage of CGM glucose values | 37.4 (4.1) | 35.5 (7.8) | 38.6 (7.8)

5. Secondary Outcome: Mean Post Prandial Excursion
Description: Difference in CGMG from the beginning of the meal challenge to the peak CGMG in the 4 hours after the meal, for both mixed meal challenges.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Insulin-only Bionic Pancreas With BC222 Lispro | Insulin-only Bionic Pancreas With Insulin Lispro | Insulin-only Bionic Pancreas With Insulin Aspart
Number analyzed (Participants) | 8 | 8 | 8
mg/dl | 95.06 (37.49) | 103.13 (47.37) | 104.07 (36.60)

6. Secondary Outcome: Number of Symptomatic Hypoglycemic Events Per Day
Description: The number of times subjects report experiencing symptoms of hypoglycemia during each bionic pancreas arm
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: number of events
Arm/Group | Insulin-only Bionic Pancreas With BC222 Lispro | Insulin-only Bionic Pancreas With Insulin Lispro | Insulin-only Bionic Pancreas With Insulin Aspart
Number analyzed (Participants) | 8 | 8 | 8
number of events | 0.73 (0.43) | 0.60 (0.43) | 1.02 (0.67)

7. Secondary Outcome: Grams of Carbohydrates Consumed to Treat Hypoglycemia Per Day
Description: The total amount of grams of carbohydrates subjects report having to take in for treatment of hypoglycemia
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: grams of carbohydrates
Arm/Group | Insulin-only Bionic Pancreas With BC222 Lispro | Insulin-only Bionic Pancreas With Insulin Lispro | Insulin-only Bionic Pancreas With Insulin Aspart
Number analyzed (Participants) | 8 | 8 | 8
grams of carbohydrates | 12.42 (11.59) | 9.27 (6.94) | 14.00 (11.95)

8. Secondary Outcome: Total Daily Dose of Insulin
Description: The average total amount of insulin delivered daily by the bionic pancreas during each bionic pancreas arm.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: units per kilogram per day
Arm/Group | Insulin-only Bionic Pancreas With BC222 Lispro | Insulin-only Bionic Pancreas With Insulin Lispro | Insulin-only Bionic Pancreas With Insulin Aspart
Number analyzed (Participants) | 8 | 8 | 8
units per kilogram per day | 0.71 (0.16) | 0.60 (0.21) | 0.61 (0.25)

ADVERSE EVENTS:
Time Frame: 1 week of study participation using each insulin, for a total of up to three weeks of study intervention
Groups:
- Insulin-only Bionic Pancreas With Insulin-aspart: Participants were randomized to complete three weeks using the insulin-only bionic pancreas. Participants would complete 7 days of each intervention in random order, including 7 days using the bionic pancreas with insulin lispro, 7 days with the bionic pancreas using insulin aspart and 7 days with the bionic pancreas using BC222 lispro. It was planned that all participants would complete all three interventions.
  The numbers listed in the participant flow, and throughout the record only represent unique participants. Dyads, including designated contacts, are not used. No data was collected from designated contacts taht is relevant to this protocol.
  The study had be terminated before all participants could complete all interventions. All available data are reported here.
Arm/Group | Insulin-only Bionic Pancreas With BC222 Lispro | Insulin-only Bionic Pancreas With Insulin Lispro | Insulin-only Bionic Pancreas With Insulin-aspart
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/9

LIMITATIONS AND CAVEATS:
The study was terminated, so only a limited number of participants completed all three interventions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/16/NCT03262116/Prot_SAP_000.pdf